CLINICAL TRIAL: NCT05516069
Title: Reaching HIV Undiagnosed: Implementation and Evaluation of Interactive Dispensing Systems for Low-barrier Access to Rapid Testing and Harm Reduction Supplies With Linkage to Care for Marginalized and Hard-to-reach Populations in Canada.
Brief Title: Our Healthbox - Evaluating Interactive Dispensing Systems for Low-Barrier Access to HIV Testing and Harm Reduction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Public Health Agency of Canada (PHAC) (Other Government); Canadian Foundation for AIDS Research (CANFAR) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-062
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: HIV; HIV Self-testing; Harm Reduction; Sexually Transmitted Diseases; Blood-Borne Infections
MeSH Terms: conditions — Harm Reduction; Sexually Transmitted Diseases; Blood-Borne Infections

STUDY DESIGN:
Intervention Model Description: Implementation science research: Cross-sectional, prospective, field trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants
  Interventions: Other: Our Healthbox (smart vending machine or interactive dispensing system)

INTERVENTIONS:
Other: Our Healthbox (smart vending machine or interactive dispensing system) — Our Healthboxes or interactive dispensing systems (IDS) will be placed in various locations across Canada and will house HIV self-test kits (provided by REACH), harm reduction supplies (provided by the provincial governments / local community based organizations; e.g. sterile drug use kits for safer injection, naloxone kits, syringes), other community determined needs (including but not limited to hats, mittens and/or socks, rapid Covid-19 antigen kits, KN95 masks). Individuals will be able to access the HIV self-test kits and harm reduction and other materials directly from the machine. Our Healthbox will also provide health information, and a support services directory for people to find the health care they need - in their community.

SUMMARY:
When REACH Nexus at MAP Centre for Urban Solutions out of St. Michael's Hospital launched its signature program, I'm Ready in 2021, our goal was to democratize access to free HIV self-testing to reach the undiagnosed in Canada. The program, the first of its kind in Canada has been successfully rolling out 50,000 free, HIV self-tests and connecting participants via a mobile app on an iOS or Android smart phone to care.

While this is an important milestone in improving access, REACH knows that more needs to be done. An estimated 20-30% of undiagnosed individuals do not have access to a phone to order the HIV self-tests, and many face multiple barriers to accessing healthcare and harm reduction support: chaotic life circumstances, addiction challenges, stigma and more.

Everyone in Canada should have equitable access to the health care they need. But REACH knows that this is not the case.So, REACH is working hard to change this. hese ongoing barriers inspired us to continue creating innovative solutions, and launch our second signature program, Our Healthbox. Our Healthbox meets people where they are, with what they need for their health and well-being. This program is scaling up innovations in health technologies to reach undiagnosed individuals with HIV. These smart interactive vending machines will be strategically located across Canada. The goal is to reach people where they live to provide free and low barrier access to HIV self-testing kits, STBBI testing and other harm reduction supplies.

Participation in Our Healthbox, as with I'm Ready, also gives us the opportunity to collect important data that will continue to inform and guide REACH Nexus' work to grow and scale innovative health solutions across the country.

DETAILED DESCRIPTION:
Our Healthbox is a national research program led by REACH Nexus part of MAP Centre for Urban Health Studies at St. Michael's Hospital, Unity Health Toronto that is rolling out "smart" vending machines across Canada. Our Healthbox provides low barrier access, connecting individuals with complex health and social needs to harm reduction materials, HIV Self-Tests and sexual health supplies.

The goal of the Our Healthbox program is to investigate whether strategically placed "smart" interactive vending machines improve access to HIV self-testing, in addition to harm reduction materials, for people who have systemic and structural barriers to accessing testing, treatment, care and prevention.

REACH Nexus is planning to launch 25-30 vending machines nationally in the first year with a goal of 100 vending machines deployed over the next 3 years. REACH is working with local community-based organizations to host and maintain the program for a minimum of 3 years.

REACH Nexus wants to reach everyone in Canada, including key populations, regardless of who they are or where they live - and to help to support them in their connection to care. There is a focus on reaching people with complex health and social needs and people who have systemic and structural barriers to accessing testing, harm reduction materials, treatment, care and prevention. Key populations include gay and bisexual men who have sex with men, African, Caribbean and Black populations, people who use substances as well as Indigenous, First Nations and Metis people.

Participants will self-recruit to the selected Our Healthbox vending machine locations. At Our Healthbox, services such as product dispensing, education information and location services information will be available to the user. Persons can view supplies and individual products to determine which items (i.e. HIV self-tests, harm reduction supplies, sexual health and wellness supplies) without registration. A location services directory is available for users to identify any nearby community based agency services near Our Healthbox.

As this is a research program, in order to dispense products (except for Naloxone for emergency use) from the machine, users will be asked to consent to the program, create a user profile and answer a few demographic questions. All information collected is anonymous, private and confidential. All products are available to the participant free of charge. For every return visit, users will sign in and answer additional survey questions prior to dispensing product. All information collected remains anonymous.

Investigators will use the RE-AIM Implementation Science Framework to outline our research objectives, questions and intended outcomes. We will evaluate if our program can:

1. reach people who are undiagnosed with HIV who have complex health, social and substance use to know their status and link to the care they need;
2. reach a significant proportion of first-time testers for HIV and subsequently link them to prevention care; and
3. provide access to harm reduction supplies to reduce harms for people who have systemic and structural barriers to accessing testing, prevention, care and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or older (except for Quebec: age 18 years or older)
* Person living in Canada (Canadian resident)
* Able to provide consent in English or French (via the machine screen)

Exclusion Criteria:

* Does not meet all inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Reaching the undiagnosed and connecting them to care | 36 months
  Number of participants who have used an HIV self test and have accessed a confirmitory HIV test (i.e. those who were undiagnosed, have tested positive for HIV and connected to care).
Reaching first time testers | 36 months
  Number of participants who report that have never tested for HIV and have accessed and used an HIV self test (i.e. first time testers).
Providing access to harm reduction supplies | 36 months
  Number of participants who access (dispense) vaious types of harm reduction supplies (e.g. injectible and non-injectible products).

CONTACTS AND LOCATIONS:
Overall Officials: Sean B Rourke, PhD, Principal Investigator — MAP Centre for Urban Health Solutions, St. Micheal's Hospital
Locations (1):
- Ensemble, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified aggregate data can be provided upon reasonbale request.

REFERENCES:
- See also: Program website — http://www.ourhealthbox.ca